CLINICAL TRIAL: NCT00228423
Title: Clopidogrel After Surgery for Coronary Artery Disease (CASCADE Trial): Does Clopidogrel Prevent Saphenous Vein Graft Disease After Coronary Bypass?
Brief Title: Trial of Clopidogrel After Surgery for Coronary Artery Disease (CASCADE Trial)
Acronym: CASCADE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Sanofi (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UOHI 2006-111
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: Atherosclerosis
Keywords: Saphenous vein; Intimal hyperplasia; Coronary artery bypass graft surgery; Antiplatelet therapy; Clopidogrel; Saphenous vein graft disease
MeSH Terms: conditions — Atherosclerosis | interventions — Clopidogrel; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 75mg Clopidogrel (Active Comparator): 75mg clopidogrel. 162mg ASA is also given, but is a standard-of-care post operative to cardiac surgery.
  Interventions: Drug: Clopidogrel 75 mg daily
- Placebo (Placebo Comparator): Water pill. 162mg ASA is also given, but is a standard-of-care post operative to cardiac surgery.
  Interventions: Drug: water pill daily

INTERVENTIONS:
Drug: Clopidogrel 75 mg daily — Daily dose of 75 mg Clopidogrel
  Arms: 75mg Clopidogrel
Drug: water pill daily — Daily dose of water pill (placebo)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the combination of clopidogrel with aspirin prevents the development of blockages (atherosclerosis) in vein grafts one year after coronary artery bypass surgery (CABG) compared to aspirin alone.

DETAILED DESCRIPTION:
Saphenous vein graft disease remains a major limitation of coronary artery bypass graft surgery (CABG). The process of saphenous vein intimal hyperplasia is mediated by platelet aggregation and begins just days after surgical revascularization. Subsequently, areas of intimal hyperplasia in turn develop graft atherosclerotic disease and its sequelae. Clopidogrel improves outcomes in patients with atherosclerotic disease, and is effective at reducing intimal hyperplasia in animal models of thrombosis. Therefore, the goal of this study will be to evaluate the efficacy of clopidogrel and aspirin therapy versus aspirin alone in the prevention of saphenous vein graft intimal hyperplasia following one year after CABG.

Patients undergoing multi-vessel CABG and in whom at least two saphenous vein grafts will be used are eligible for the study. Patients will be randomized to receive daily clopidogrel 75 mg or placebo, in addition to daily aspirin 162 mg, for the duration of one year starting as soon as postoperative bleeding has been ruled out on the day of surgery. At the end of one year, all patients will undergo coronary angiography and intravascular ultrasound assessment of one saphenous vein graft as selected by randomization. The study will be powered to test the hypothesis that clopidogrel and aspirin will reduce vein graft intimal hyperplasia by 20% compared to aspirin alone at one year following bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary multi-vessel CABG with at least two saphenous vein grafts, with or without the use of cardiopulmonary bypass.

Exclusion Criteria:

* Emergency surgery
* Valve surgery
* Redo CABG
* Left ventricle ejection fraction < 25%
* Serum creatinine > 130 µmol/L
* Preoperative use of clopidogrel (with the exception of the current admission)
* Preoperative use of warfarin; allergy to aspirin or clopidogrel.
* History of cerebrovascular accident
* History of severe liver disease
* Morbid obesity
* Current malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2006-05; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ruel, MD, MPH, Principal Investigator — Ottawa Heart Institute Research Corporation; Alexander Kulik, MD, Study Director — Ottawa Heart Institute Research Corporation; Michel Le May, MD, Study Director — Ottawa Heart Institute Research Corporation; George A Wells, PhD, Study Director — Ottawa Heart Institute Research Corporation; Thierry G Mesana, MD, PhD, Study Director — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Fitzgibbon GM, Kafka HP, Leach AJ, Keon WJ, Hooper GD, Burton JR. Coronary bypass graft fate and patient outcome: angiographic follow-up of 5,065 grafts related to survival and reoperation in 1,388 patients during 25 years. J Am Coll Cardiol. 1996 Sep;28(3):616-26. doi: 10.1016/0735-1097(96)00206-9. PMID 8772748
- [Background] Motwani JG, Topol EJ. Aortocoronary saphenous vein graft disease: pathogenesis, predisposition, and prevention. Circulation. 1998 Mar 10;97(9):916-31. doi: 10.1161/01.cir.97.9.916. PMID 9521341
- [Background] Jawien A, Bowen-Pope DF, Lindner V, Schwartz SM, Clowes AW. Platelet-derived growth factor promotes smooth muscle migration and intimal thickening in a rat model of balloon angioplasty. J Clin Invest. 1992 Feb;89(2):507-11. doi: 10.1172/JCI115613. PMID 1531345
- [Background] Herbert JM, Dol F, Bernat A, Falotico R, Lale A, Savi P. The antiaggregating and antithrombotic activity of clopidogrel is potentiated by aspirin in several experimental models in the rabbit. Thromb Haemost. 1998 Sep;80(3):512-8. PMID 9759636
- [Background] Herbert JM, Tissinier A, Defreyn G, Maffrand JP. Inhibitory effect of clopidogrel on platelet adhesion and intimal proliferation after arterial injury in rabbits. Arterioscler Thromb. 1993 Aug;13(8):1171-9. doi: 10.1161/01.atv.13.8.1171. PMID 8343491
- [Background] Hermann A, Weber AA, Schror K. Clopidogrel inhibits platelet adhesion and platelet-dependent mitogenesis in vascular smooth muscle cells. Thromb Res. 2002 Jan 15;105(2):173-5. doi: 10.1016/s0049-3848(01)00403-0. No abstract available. PMID 11958809
- [Background] Harker LA, Marzec UM, Kelly AB, Chronos NR, Sundell IB, Hanson SR, Herbert JM. Clopidogrel inhibition of stent, graft, and vascular thrombogenesis with antithrombotic enhancement by aspirin in nonhuman primates. Circulation. 1998 Dec 1;98(22):2461-9. doi: 10.1161/01.cir.98.22.2461. PMID 9832493
- [Background] Cadroy Y, Bossavy JP, Thalamas C, Sagnard L, Sakariassen K, Boneu B. Early potent antithrombotic effect with combined aspirin and a loading dose of clopidogrel on experimental arterial thrombogenesis in humans. Circulation. 2000 Jun 20;101(24):2823-8. doi: 10.1161/01.cir.101.24.2823. PMID 10859288
- [Background] Bhatt DL, Chew DP, Hirsch AT, Ringleb PA, Hacke W, Topol EJ. Superiority of clopidogrel versus aspirin in patients with prior cardiac surgery. Circulation. 2001 Jan 23;103(3):363-8. doi: 10.1161/01.cir.103.3.363. PMID 11157686
- [Background] Fox KA, Mehta SR, Peters R, Zhao F, Lakkis N, Gersh BJ, Yusuf S; Clopidogrel in Unstable angina to prevent Recurrent ischemic Events Trial. Benefits and risks of the combination of clopidogrel and aspirin in patients undergoing surgical revascularization for non-ST-elevation acute coronary syndrome: the Clopidogrel in Unstable angina to prevent Recurrent ischemic Events (CURE) Trial. Circulation. 2004 Sep 7;110(10):1202-8. doi: 10.1161/01.CIR.0000140675.85342.1B. Epub 2004 Aug 16. PMID 15313956
- [Result] Kulik A, Le May M, Wells GA, Mesana TG, Ruel M. The clopidogrel after surgery for coronary artery disease (CASCADE) randomized controlled trial: clopidogrel and aspirin versus aspirin alone after coronary bypass surgery [NCT00228423]. Curr Control Trials Cardiovasc Med. 2005 Oct 11;6(1):15. doi: 10.1186/1468-6708-6-15. PMID 16219100
- [Result] Kulik A, Le May MR, Voisine P, Tardif JC, Delarochelliere R, Naidoo S, Wells GA, Mesana TG, Ruel M. Aspirin plus clopidogrel versus aspirin alone after coronary artery bypass grafting: the clopidogrel after surgery for coronary artery disease (CASCADE) Trial. Circulation. 2010 Dec 21;122(25):2680-7. doi: 10.1161/CIRCULATIONAHA.110.978007. Epub 2010 Dec 6. PMID 21135365
- [Result] Kulik A, Voisine P, Mathieu P, Masters RG, Mesana TG, Le May MR, Ruel M. Statin therapy and saphenous vein graft disease after coronary bypass surgery: analysis from the CASCADE randomized trial. Ann Thorac Surg. 2011 Oct;92(4):1284-90; discussion 1290-1. doi: 10.1016/j.athoracsur.2011.04.107. PMID 21958773
- [Result] Une D, Kulik A, Voisine P, Le May M, Ruel M. Correlates of saphenous vein graft hyperplasia and occlusion 1 year after coronary artery bypass grafting: analysis from the CASCADE randomized trial. Circulation. 2013 Sep 10;128(11 Suppl 1):S213-8. doi: 10.1161/CIRCULATIONAHA.112.000328. PMID 24030409
- [Result] Une D, Al-Atassi T, Kulik A, Voisine P, Le May M, Ruel M. Impact of clopidogrel plus aspirin versus aspirin alone on the progression of native coronary artery disease after bypass surgery: analysis from the Clopidogrel After Surgery for Coronary Artery DiseasE (CASCADE) randomized trial. Circulation. 2014 Sep 9;130(11 Suppl 1):S12-8. doi: 10.1161/CIRCULATIONAHA.113.008227. PMID 25200049
- [Derived] Hage A, Voisine P, Erthal F, Larose E, Glineur D, Chow B, Tremblay H, Fortier J, Ko G, Une D, Farkouh M, Mesana TG, LeMay M, Kulik A, Ruel M. Eight-year follow-up of the Clopidogrel After Surgery for Coronary Artery Disease (CASCADE) trial. J Thorac Cardiovasc Surg. 2018 Jan;155(1):212-222.e2. doi: 10.1016/j.jtcvs.2017.06.039. Epub 2017 Jun 24. PMID 28734623
- See also: University of Ottawa Heart Institute Website — http://www.ottawaheart.ca/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 75mg Clopidogrel | Placebo
Started | 56 | 57
Completed | 46 | 45
Not Completed | 10 | 12
Not completed — Adverse Event | 2 | 5
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Protocol Violation | 1 | 3
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 75mg Clopidogrel | Placebo | Total
Number analyzed (Participants) | 56 | 57 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (7.5) | 68.1 (7.4) | 66.0 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 51 | 50 | 101

OUTCOME MEASURES:

1. Primary Outcome: Vein Graft Intimal Area
Description: IVUS imaging 12 months post-CABG, and the average intimal area in the proximal 40 mm of one vein graft per patient will be assessed
Time Frame: One year following surgery
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 75mg Clopidogrel | Placebo
Number analyzed (Participants) | 46 | 44
mm | 4.1 (2.0) | 4.5 (2.1)

2. Secondary Outcome: Vein Graft Angiographic Patency
Description: Postoperative angiogram 12 months post-CABG
Time Frame: One year following surgery
Measure: Number; unit: percentage
Arm/Group | 75mg Clopidogrel | Placebo
Number analyzed (Participants) | 46 | 44
percentage | 94.3 | 93.2

3. Secondary Outcome: Incidence of Major Adverse Coronary Events Within One Year Following Surgery
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 75mg Clopidogrel | Placebo
Number analyzed (Participants) | 56 | 57
Participants | 4 | 5

4. Secondary Outcome: Incidence of Major Bleeding Events Within One Year Following Surgery
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 75mg Clopidogrel | Placebo
Number analyzed (Participants) | 56 | 57
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 75mg Clopidogrel | Placebo
All-Cause Mortality (participants affected / at risk) | 0/56 | 1/57
Serious Adverse Events (participants affected / at risk) | 4/56 | 5/57
Other Adverse Events (participants affected / at risk) | 3/56 | 3/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 75mg Clopidogrel (N=56) | Placebo (N=57)
Myocardial infarction (Cardiac disorders) | 4 (4) | 0 (0)
Cerebrovascular accident (Cardiac disorders) | 0 (0) | 2 (2)
Hospitalization for Coronary Ischemia (Cardiac disorders) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 75mg Clopidogrel (N=56) | Placebo (N=57)
Minor bleeding (General disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication will be a joint effort between all contributing parties. At least 30 days before submission for publication, the partnership will be provided the proposed publication and will be given 30 days to respond with approval or requests for holds. All contributing parties must be acknowledged in all publications.